CLINICAL TRIAL: NCT03532919
Title: Heart and Renal Failure in Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bengt Nellgard, Associate professor, Sahlgrenska University Hospital
Other Study IDs: Refhina
Record Dates: First submitted 2018-04-10; First posted 2018-05-22 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Hypotension; Hip Fractures; Renal Insufficiency; Heart Injuries
MeSH Terms: conditions — Hypotension; Hip Fractures; Renal Insufficiency; Heart Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Laboratory samples on Creatinin Cystatin C NTproBNP and Troponin T
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum Tropinin — Blodsamples will be taken 4 times from preoperatively to 2 Days postoperatively
  Other Names: Serum Cystatin C

SUMMARY:
Patients with acute hip fractures are old and vulnerable. With a majoriry classified as being ASA 3 or more. Frequently they receive spinal anesthesia perioperatively inducing hypotension. Even a short hypotensive period may induce postop cardiac T roponinT leakage as well as renal failure noted by Changes in Serum Creatinin or Cýstatin C This will be investigated and correlated to intraoperative hypotension as step one. Preliminary this will be followed by an intervention with vasopressor treatment perioperatively to preserve an adequte MABP

DETAILED DESCRIPTION:
Patients with acute hip fractures are old and vulnerable. With a majoriry classified as being ASA 3 or more. Frequently they receive spinal anesthesia perioperatively inducing hypotension. Even a short hypotensive period may induce postop cardiac T roponinT leakage as awell as renal failure noted by Changes in S Creatinin or Cýstatin C This will be investigated and correlated to intraoperative hypotension as a step one. Preliminary this will be followed by an intervention with vasopressor treatment perioperatively to preserve an adequte MABP

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture patient to be operated upon Classified as being ASA 3 or more

Exclusion Criteria:

* Not forfilling inclusion Criterias

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an acute hip fracture classified as being ASA 3 or more
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days
  post surgery

SECONDARY OUTCOMES:
Serum concentrations of Troponin, NTproBNP, Creatinin and Cystatin C | 90 days
  Relations between values and mortality at 30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bengt M Nellgard, MD PhD, Principal Investigator — SahlgrenskaUniversity Hospital
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided